CLINICAL TRIAL: NCT04316871
Title: Epidural Morphine for Geriatrics Undergoing Lower Abdominal Cancer Surgery: a Dose Response Study
Brief Title: Dosage of Epidural Morphine in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Muhammad Mostafa Shawqi Abdelnasser, Anesthesia resident at South Egypt Cancer Institute, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EPMDose
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Age Problem; Abdominal Cancer
Keywords: Injections, Epidural; Morphine Sulfate
MeSH Terms: interventions — Morphine; Saline Solution; Fumigant 93

STUDY DESIGN:
Intervention Model Description: This randomized, double blinded, clinical trial was approved by the local ethics committee of faculty of medicine, Assuit University, Assuit, Egypt. The maximum total PCA morphine consumption was 12 ± 16 mg while in healthy controls was 70± 35 mg. We aim to enroll at least 60-80 participants considering the following assumptions:
  * Main statistical test is ANOVA\t-test to detect the difference of the difference of PCA morphine consumption between the four groups.
  * Main outcome variable is total PCA morphine consumption after lower abdominal cancer surgery in elderly patients receiving three different doses of epidural morphine in comparison with its consumption in healthy controls not receiving epidural morphine.
  * Effect size = 0.75, Alpha = 0.05, Power = 0.80
  * Allocation ratio N4/N3/N2/N1 = 1/1/1/1.
  * 22 patients should be enrolled in each group to account for dropouts.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group D (Placebo Comparator): A total volume of 10 mL injection 5 mL of bupivacaine hydrochloride 0.125% diluted in 5 mL preservative-free normal saline by the hospital pharmacist.
  Interventions: Drug: Normal saline
- Group A (Active Comparator): A total volume of 10 mL injection: 5 mL of bupivacaine hydrochloride 0.125% with 1.5 mg of preservative-free morphine diluted in 5 mL preservative-free normal saline by the hospital pharmacist.
  Interventions: Drug: 1.5 mg of Morphine Sulfate
- Group B (Active Comparator): A total volume of 10 mL injection: 5 mL of bupivacaine hydrochloride 0.125% with 3 mg of preservative-free morphine diluted in 5 mL preservative-free normal saline by the hospital pharmacist.
  Interventions: Drug: 3 mg of Morphine Sulfate
- Group C (Active Comparator): A total volume of 10 mL injection: 5 mL of bupivacaine hydrochloride 0.125% with 4 mg of preservative-free morphine diluted in 5 mL preservative-free normal saline by the hospital pharmacist.
  Interventions: Drug: 4.5 mg of Morphine Sulfate

INTERVENTIONS:
Drug: 1.5 mg of Morphine Sulfate — 1.5 mg of Morphine Sulphate will be given epidurally.
  Other Names: A
  Arms: Group A
Drug: Normal saline — Normal saline will be given epidurally.
  Other Names: D
  Arms: Group D
Drug: 3 mg of Morphine Sulfate — 3 mg of Morphine Sulphate will be given epidurally.
  Other Names: B
  Arms: Group B
Drug: 4.5 mg of Morphine Sulfate — 4.5 mg of Morphine Sulphate will be given epidurally.
  Other Names: C
  Arms: Group C

SUMMARY:
This a clinical trial that evaluates the efficacy and safety of three different doses of morphine, namely 1.5 mg, 3 mg and 4.5 mg, via the epidural route regarding reducing pain in elderly patients after a cancer surgery in the lower abdomen

DETAILED DESCRIPTION:
Acute postoperative pain is a common complaint for several days after surgery. However, acute postoperative pain remains even more under controlled in elderly patients, especially those with cognitive impairment and malignancy. Geriatric population is reported to be at higher risk for unwanted side effects from analgesic treatments compared to younger patients due to different major risk factors such as: decline in organ function, polypharmacy, pharmacokinetics, drug sensitivity, and frailty. Despite of the higher risk of opioids, especially morphine, causing toxicity and adverse effect; they are still the cornerstone treatment of severe acute postoperative pain. Morphine in those patients is very likely to cause toxicity because of accumulation of its active metabolites compared to other opioids with fewer or no active metabolites. Epidural morphine is an effective route for an effective drug. Furthermore, unwanted side effects with neuraxial opioids are minor and managed easily. Regarding clinical outcomes, clinical studies showed a lot of improvements associated with postoperative opioid analgesia. Now, there is a clinical necessity to achieve the best management of acute postoperative pain in elderly patients with the least possibility of adverse side effects. We aim in this randomized, assessor blinded, clinical trial at Assuit University to determine the optimum dose of epidural morphine for the highest control of acute postoperative pain in geriatrics who are planned to have lower abdominal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥ 60 years, who are planned to undergo lower abdominal cancer surgery.

2- ASA I and II classifications. 2. Surgeries via infra-umbilical abdominal incision is considered eligible.

Exclusion Criteria:

1. Patient refusal.
2. Patients who are morbidly obese (body mass index ≥ 40 kg/m2).
3. Those with contraindications to neuraxial analgesia. 4- psychiatric illness that would interfere with the perception and the assessment of pain.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diab Hetta, MD, Study Director — Assiut University
Locations (1):
- Assuit University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study will be available from the corresponding author on reasonable request. The data will not be publicly available due to containing information that could compromise research participant privacy/consent.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will not be publicly available due to containing information that could compromise research participant privacy/consent.
Access Criteria: The data will not be publicly available due to containing information that could compromise research participant privacy/consent.

REFERENCES:
- [Background] McKeown JL. Pain Management Issues for the Geriatric Surgical Patient. Anesthesiol Clin. 2015 Sep;33(3):563-76. doi: 10.1016/j.anclin.2015.05.010. Epub 2015 Jul 3. PMID 26315638
- [Background] Palmer CM, Nogami WM, Van Maren G, Alves DM. Postcesarean epidural morphine: a dose-response study. Anesth Analg. 2000 Apr;90(4):887-91. doi: 10.1097/00000539-200004000-00021. PMID 10735794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at South Egypt Cancer institute and Assiut university hospitals according to Consolidated Standards of Reporting Trials (CONSORT) statement. Patients were recruited from the departments of surgical oncology between March 2020 and June 2021.
Pre-assignment Details: A total of 102 patients were assessed for eligibility. Three of them refused to participate in the study, and three did not meet the inclusion criteria.
Groups:
- Group A (1.5 mg): Participants were allocated to receive epidural morphine 1.5 mg group.
- Group B (3 mg): Participants were allocated to receive epidural morphine 3 mg group.
- Group C (4.5mg): Participants were allocated to receive epidural morphine 4.5 mg group.
- Group D (0 mg): Participants were allocated to receive epidural morphine 0 mg group.
Period: Overall Study
Arm/Group | Group A (1.5 mg) | Group B (3 mg) | Group C (4.5mg) | Group D (0 mg)
Started | 24 | 24 | 24 | 24
Completed | 22 | 22 | 22 | 22
Not Completed | 2 | 2 | 2 | 2
Not completed — Protocol Violation | 2 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Incomplete data of eight participants was excluded from the final analysis due to protocol violation.
Groups:
- Group A: Participants allocated to receive 1.5 mg epidural morphine.
- Group B: Participants allocated to receive 3 mg epidural morphine.
- Group C: Participants allocated to receive 4.5 mg epidural morphine.
- Group D: Participants allocated to receive 0 mg epidural morphine.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Incomplete data of eight participants was excluded from the final analysis due to protocol violation. In group D, one was excluded due to failed epidural, and the other was excluded due to erroneous intake of IV fentanyl. In group A, one was excluded due to failed epidural, and the other was excluded due to unresectable tumor. In group B, one was excluded due to failed epidural, and the other patient was excluded due to redo of surgery. In group C, two were excluded due to failed epidural.
  Years | 66.82 (7.500) | 65.32 (5.498) | 65.27 (5.373) | 64.32 (4.145) | 65.43 (5.629)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Incomplete data of eight participants was excluded from the final analysis due to protocol violation. In group D, one was excluded due to failed epidural, and the other was excluded due to erroneous intake of IV fentanyl. In group A, one was excluded due to failed epidural, and the other was excluded due to unresectable tumor. In group B, one was excluded due to failed epidural, and the other patient was excluded due to redo of surgery. In group C, two were excluded due to failed epidural.
  Participants
    Female | 14 | 16 | 12 | 15 | 57
    Male | 8 | 6 | 10 | 7 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Incomplete data of eight participants was excluded from the final analysis due to protocol violation. In group D, one was excluded due to failed epidural, and the other was excluded due to erroneous intake of IV fentanyl. In group A, one was excluded due to failed epidural, and the other was excluded due to unresectable tumor. In group B, one was excluded due to failed epidural, and the other patient was excluded due to redo of surgery. In group C, two were excluded due to failed epidural.
  Participants
    Egyptian Population | 22 | 22 | 22 | 22 | 88
Region of Enrollment [Number; unit: participants] — Population: Incomplete data of eight participants was excluded from the final analysis due to protocol violation. In group D, one was excluded due to failed epidural, and the other was excluded due to erroneous intake of IV fentanyl. In group A, one was excluded due to failed epidural, and the other was excluded due to unresectable tumor. In group B, one was excluded due to failed epidural, and the other patient was excluded due to redo of surgery. In group C, two were excluded due to failed epidural.
  participants
    Egypt | 22 | 22 | 22 | 22 | 88
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Incomplete data of eight participants was excluded from the final analysis due to protocol violation. In group D, one was excluded due to failed epidural, and the other was excluded due to erroneous intake of IV fentanyl. In group A, one was excluded due to failed epidural, and the other was excluded due to unresectable tumor. In group B, one was excluded due to failed epidural, and the other patient was excluded due to redo of surgery. In group C, two were excluded due to failed epidural.
  kg/m^2 | 25 (3.423) | 26.18 (3.202) | 24.59 (4.148) | 26.18 (3.711) | 25.49 (3.621)

OUTCOME MEASURES:

1. Primary Outcome: Total Patient-controlled Analgesia (PCA) Morphine Sulphate (MS) Consumption.
Description: The mean total PCA morphine consumption (mg) in the first 72 hr. postoperatively
Time Frame: 72 hours
Population: Main statistical test is ANOVA\t-test to detect the difference of PCA morphine consumption between the four groups.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 22 | 22 | 22 | 22
mg | 27.182 (5.6115) | 9.182 (3.5273) | 6.273 (3.4307) | 38.136 (4.8037)

2. Secondary Outcome: Visual Analog Scale
Description: Visual Analog Scale is a visual chart scored from 0 (no pain) to 10 ( the worst pain ever) used by the patient to report the severity of their pain to assess the pain intensity, and all patients were instructed how to evaluate their pain and how to use the patient-controlled analgesia.
Time Frame: 72 hours
Population: Main statistical test is ANOVA\t-test to detect the difference of between the four groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 22 | 22 | 22 | 22
units on a scale | 3.95 (1.09) | 2.00 (0.756) | 1.68 (1.041) | 4.32 (1.129)

3. Secondary Outcome: Modified Ramsay Sedation Scale
Description: It is an six-point scale informed by degree of responsiveness to verbal and tactile stimulus where awake levels were as follows:
  I = anxious, agitated, or restless; II = cooperative, oriented, and tranquil; III = response to command, and asleep levels were dependent on the patient's response to a light glabellar tap or loud auditory stimulus; IV = brisk response; V = a sluggish response; and VI = no response
Time Frame: Modified Ramsay Sedation Scale at 2 hours postoperative
Population: Main statistical test is ANOVA\t-test to detect the difference between the four groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 22 | 22 | 22 | 22
score on a scale | 1.95 (0.375) | 2.18 (0.395) | 3.05 (0.375) | 1.86 (0.468)

4. Secondary Outcome: Nausea Score
Description: It is a subjective scale to assess the nauseating side effects of morphine at eight time points (0, 2, 8, 16, 24, 36, 48 and 72 h). The 72-hour score for this side effect was the sum of these eight scores. Nausea scores were recorded on a scale with a minimum of 0 to a maximum of 2; where:
  0 was recorded if the side effect was absent;
  1. if the side effect was minimal and did not require treatment;
  2. if the side effect was moderate or severe and required treatment.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 22 | 22 | 22 | 22
scores on a scale | 4.41 (0.796) | 4.45 (0.739) | 4.59 (0.734) | 4.82 (0.733)

5. Secondary Outcome: Vomiting Score
Description: It is a subjective scale to assess the vomiting as a side effect of epidural morphine at eight time points (0, 2, 8, 16, 24, 36, 48 and 72 h). The 72-hour score for this side effect was the sum of these eight scores. Vomiting scores were recorded on a scale with a minimum of 0 to a maximum of 2; where:
  0 was recorded if the side effect was absent;
  1. if the side effect was minimal and did not require treatment;
  2. if the side effect was moderate or severe and required treatment.
Time Frame: 72 hours
Population: Main statistical test is ANOVA\t-test to detect the difference of between the four groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 22 | 22 | 22 | 22
score on a scale | 3.18 (0.958) | 3.00 (1.902) | 3.86 (2.122) | 1.45 (1.224)

6. Secondary Outcome: Pruritus Score
Description: It is a subjective scale to assess the pruritus as a side effect of morphine at eight time points (0, 2, 8, 16, 24, 36, 48 and 72 h). The 72-hour score for this side effect was the sum of these eight scores. Pruritus scores were recorded on a scale with a minimum of 0 to a maximum of 2; where:
  0 was recorded if the side effect was absent;
  1. if the side effect was minimal and did not require treatment;
  2. if the side effect was moderate or severe and required treatment.
Time Frame: 72 hours
Population: Main statistical test is ANOVA\t-test to detect the difference of between the four groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 22 | 22 | 22 | 22
score on a scale | 3.36 (0.953) | 3.68 (1.086) | 3.23 (0.752) | 1.91 (1.377)

ADVERSE EVENTS:
Time Frame: 72 hours
Description: Postoperative sedation effect of epidural morphine was frequently assessed by Modified Ramsay sedation scale. All-Cause Mortality and serious adverse events were not monitored/assessed.
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 1/22 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=22) | Group B (N=22) | Group C (N=22) | Group D (N=22)
Modified Ramsay Sedation Score; level V (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) — sluggish response.

LIMITATIONS AND CAVEATS:
This study is limited by focusing on lower abdominal cancer surgeries only; also, it is a single center study. Therefore, the generalizability of our results is limited. Future large studies on different types of surgeries are needed. Due to the vulnerability of older adults, we assessed the balancing dose of epidural morphine versus age only. The relation between the dose of epidural morphine and common comorbidities in this age group should be investigated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT04316871/Prot_SAP_000.pdf